CLINICAL TRIAL: NCT00057876
Title: A Randomized Phase III Study Of Gemcitabine In Combination With Radiation Therapy Versus Gemcitabine Alone In Patients With Localized, Unresectable Pancreatic Cancer
Brief Title: Gemcitabine With or Without Radiation Therapy in Treating Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000278947; U10CA021115 (NIH); E4201 (Other: Eastern Cooperative Oncology Group (ECOG) and Radiation Therapy Oncology Group (RTOG))
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine (Active Comparator)
  Interventions: Drug: Gemcitabine
- Gemcitabine + Radiation (Experimental)
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Drug: Gemcitabine — Induction: Patients receive the first cycle of gemcitabine 1000 mg/m^2 intravenously once per week for 6 weeks followed by 1 week rest.
  Consolidation: Following the week of rest, treatment resume with gemcitabine 1000 mg/m^2 administered intravenously once per week for 3 weeks, followed by 1 week rest, for 5 (4-week) cycles.
  Other Names: 2-Deoxy-2; 2-difluorocytidine monohydrochloride; Gemzar
  Arms: Gemcitabine
Radiation: radiation therapy — Induction: Patients receive gemcitabine 600 mg/m^2 intravenous infusion over 30-60 minutes once a week for 6 weeks while receiving radiation therapy. The first gemcitabine dose is given on the first day of radiation therapy (prior to radiation), then weekly thereafter. All patients on Arm B receive radiation therapy Monday through Friday (no radiation on Saturday or Sunday), weeks 1-6, with once/week gemcitabine. The radiation dose per fraction is 180 cGy prescribed to the isocenter. The total dose of radiation is 5040 cGy given in 28 fractions over 5 1/2 weeks.
  Consolidation: Additional cycles of gemcitabine begin approximately 4 weeks after completion of radiation therapy.
  Other Names: 2-Deoxy-2; 2-difluorocytidine monohydrochloride; Gemzar
  Arms: Gemcitabine + Radiation

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether gemcitabine is more effective with or without radiation therapy in treating pancreatic cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of gemcitabine with or without radiation therapy in treating patients who have locally advanced, unresectable pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and progression-free of patients with locally advanced, unresectable pancreatic cancer treated with gemcitabine with or without radiotherapy.
* Compare the objective response rate in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life (QOL) of patients treated with these regimens.
* Determine the effect of gemcitabine and radiotherapy on the QOL of patients with improved objective response rate and progression-free and overall survival.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to performance status (0 vs. 1) and weight loss within the past 6 months (less than 10% vs. 10% or more). Patients are randomized to 1 of 2 treatment arms.

Arm I (Gemcitabine alone):

* Induction: Patients receive gemcitabine intravenously (IV) over 30-60 minutes once weekly for 6 weeks followed by 1 week of rest.
* Consolidation: After the 1 week of rest, patients receive gemcitabine IV once weekly for 3 weeks. Treatment repeats every 4 weeks for 5 courses in the absence of disease progression or unacceptable toxicity.

Arm II (Gemcitabine with radiotherapy):

* Induction: Patients receive gemcitabine IV over 30-60 minutes once weekly for 6 weeks beginning on day 1. Patients also undergo concurrent radiotherapy 5 days a week for 5.5 weeks beginning on day 1.
* Consolidation: Approximately 4 weeks after completion of radiotherapy, patients receive gemcitabine IV over 30-60 minutes once weekly for 3 weeks. Treatment repeats every 4 weeks for 5 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, week 6, week 15 (for arm II), week 16 (for arm I), and 9 months.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year. Patients who receive treatment beyond 3 years are followed for survival.

ACCRUAL: 74 patients were accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Locally advanced or regional (encompassable within the same radiotherapy portals)
  * Adenosquamous cancers are allowed
* Unresectable disease
* Measurable and/or non-measurable disease as determined by computed tomography (CT) scan or magnetic resonance imaging (MRI), which must be performed within 4 weeks prior to randomization.
* Age>=18
* ECOG Performance status of 0-1
* Life expectancy >= 12 weeks
* Adequate bone marrow reserve,liver and renal function within 2 weeks of randomization:

  * Absolute granulocyte count at least 2,000/mm^3
  * Platelet count at least 100,000/mm^3
  * Bilirubin less than 3 mg/dL (unless secondary to biliary obstruction or cholangitis)
  * Serum glutamic-oxaloacetic (AST) less than 5 times upper limit of normal (ULN)
  * Albumin greater than 2.5 g/dL
  * Creatinine no greater than 1.5 times ULN
* Fertile patients must use effective contraception
* Willing and able to attend follow-up visits
* Concurrent enrollment on protocol ECOG-E1Y03 allowed
* More than 4 weeks since prior investigational agents

Exclusion Criteria:

* Candidate for surgical excision based on local extent of disease (e.g., T3, N1, M0)
* Stage M1 disease
* Small cell, mucinous cystadenocarcinoma, islet cell or papillary cystic histology
* Pregnant or nursing
* Active infection within within 4 weeks of randomization
* Malignancy within the past 5 years except nonmelanoma skin cancer, carcinoma in situ of the cervix, or organ-confined prostate cancer (Gleason score no greater than 7)
* History of active collagen vascular disease (i.e., systemic lupus erythematosus, rheumatoid arthritis, or scleroderma)
* Signs or symptoms of peptic or duodenal ulcer disease
* Concurrent serious systemic disorders that are incompatible with study participation
* Prior chemotherapy for pancreatic cancer
* Prior radiotherapy
* Concurrent intensity modulated radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2003-08-29 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Loehrer, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (229):
- United States (228):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Saint Joseph's Mercy Cancer Center, Hot Springs, Arkansas
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Doctors Medical Center, Modesto, California
  - Memorial Medical Center Cancer Services, Modesto, California
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - New Britain General Hospital, New Britain, Connecticut
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - William W. Backus Hospital, Norwich, Connecticut
  - Halifax Medical Center, Daytona Beach, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Cancer Care and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Wasser Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Deerpath Medical Associates, Lake Forest, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Northwest Medical Specialist, PC, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates at June E. Nylen Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Good Samaritan Health Systems, Kearney, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Shore Memorial Hospital - Somers Point, Somers Point, New Jersey
  - Community Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Louis Busch Hager Cancer Center at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - St. Elizabeth Boardman Cancer Center, Boardman, Ohio
  - University Hospitals Ireland Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - St. Joseph Health Care Center, Warren, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - St. Elizabeth Cancer Center at St. Elizabeth Health Center - Youngstown, Youngstown, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Center - Sayre, Sayre, Pennsylvania
  - Hematology and Oncology Associates, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, P. C., Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baptist Regional Cancer Center at Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - East Texas Medical Center Cancer Institute, Tyler, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Bon Secours Cancer Care at St. Mary's Hospital, Richmond, Virginia
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Marshall University Medical Center, Huntington, West Virginia
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Cancer Care Center at Holy Family Memorial Medical Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconsin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Loehrer PJ, Powell ME, Cardenes HR, et al.: A randomized phase III study of gemcitabine in combination with radiation therapy versus gemcitabine alone in patients with localized, unresectable pancreatic cancer: E4201. [Abstract] J Clin Oncol 26 (Suppl 15): A-4506, 2008.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on April 10,2003, accrued its first patient on August 29, 2003, and terminated on December 15, 2005 as a result of slow accrual. The final accrual of the study was 74 patients. This was an intergroup study and coordinated by Eastern Cooperative Oncology Group with 9 participating groups.
Groups:
- Gemcitabine: Induction: Patients will receive the first cycle of gemcitabine 1000 mg/m² intravenously once per week for 6 weeks followed by 1 week rest.
  Consolidation: Following the week of rest, treatment will resume with 1000 mg/m² administered intravenously once per week for 3 weeks, followed by 1 week rest, for 5 (4-week) cycles.
- Gemcitabine + Radiation: Induction: Patients will receive gemcitabine 600 mg/m² intravenous infusion over 30-60 minutes once a week for 6 weeks while receiving radiation therapy. The first gemcitabine dose will be given on the first day of radiation therapy (prior to radiation), then weekly thereafter. All patients on Arm B will receive radiation therapy Monday through Friday (no radiation on Saturday or Sunday), weeks 1-6, with once/week gemcitabine. The radiation dose per fraction will be 180 cGy prescribed to the isocenter. The total dose of radiation will be 5040 cGy given in 28 fractions over 5 1/2 weeks.
  Consolidation: Additional cycles of gemcitabine will begin approximately 4 weeks after completion of radiation therapy.
Period: Overall Study
Arm/Group | Gemcitabine | Gemcitabine + Radiation
Started | 38 | 36
Eligible | 37 | 34
Began Protocol Therapy | 35 | 34
Eligible and Treated | 34 | 34
Completed | 9 | 9
Not Completed | 29 | 27
Not completed — Adverse Event | 8 | 8
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lack of Efficacy | 10 | 8
Not completed — Ineligible | 1 | 2
Not completed — other reason | 2 | 2
Not completed — other complicating disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine | Gemcitabine + Radiation | Total
Number analyzed (Participants) | 37 | 34 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (8.7) | 65.3 (10.3) | 66.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 18 | 19 | 37
Region of Enrollment [Number; unit: participants]
  United States | 37 | 34 | 71

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time
Description: Overall survival was defined as the time from randomization (registration) to death from any cause. Patients alive at last follow-up were censored. Patients were followed every 3 months for 2 years and then every 6 months for year 3. Patients received treatment beyond 3 years were also followed for survival.
Time Frame: assessed every 3 months for 2 years, then every 6 months for year 3
Population: 71 eligible patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine | Gemcitabine + Radiation
Number analyzed (Participants) | 37 | 34
Months | 9.2 [7.9 to 11.4] | 11.0 [7.6 to 15.5]
Statistical Analysis 1: Comparison: Gemcitabine vs Gemcitabine + Radiation; Log rank test is conducted for OS to see whether the two treatment arms are different in their overall survival probabilities; Test type: Superiority or Other; p = 0.017, Log Rank

2. Secondary Outcome: Progression-free Survival Time
Description: Time from randomization (registration) to the earlier of disease progression or death. Patients alive and progression-free at last follow-up were censored. Progressive disease was defined as at least a 20% increase in the sum of the longest diameters of target lesions (taking as reference the baseline sum longest diameter), or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Patients were followed every 3 months for 2 years and then every 6 months for year 3. Patients who received treatment beyond 3 years were also followed for survival.
Time Frame: assessed every 3 months for 2 years, then every 6 months for year 3
Population: 67 eligible patients with data on progression-free survival(PFS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine | Gemcitabine + Radiation
Number analyzed (Participants) | 34 | 33
Months | 6.7 [3.9 to 8.7] | 6.0 [5.4 to 8.4]
Statistical Analysis 1: Comparison: Gemcitabine vs Gemcitabine + Radiation; Test type: Superiority or Other; p = 0.25, Log Rank

3. Secondary Outcome: Overall Response
Description: Response was assessed per Response Evaluation Criteria In Solid Tumors (RECIST) by CT. Overall response included complete response (CR) and partial response (PR). CR was defined as the disappearance of all target and non-target lesions. PR was defined as CR of target lesions and persistence of one or more non-target lesions or at least a 30% decrease in the sum of the longest diameters of target lesions and non-progressive disease in the non-target lesions. The 71 eligible, treated participants were included in the analysis.
Time Frame: assessed at week 8, and every 3 months for 2 years, then every 6 months for year 3
Population: Eligible patients
Measure: Number; unit: participants
Arm/Group | Gemcitabine | Gemcitabine + Radiation
Number analyzed (Participants) | 37 | 34
participants | 2 | 2
Statistical Analysis 1: Comparison: Gemcitabine vs Gemcitabine + Radiation; Compare objective response rate (CR+PR) between two treatment groups; Test type: Superiority or Other; p = 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: Assessed at the end of the rest period following induction, and again 4 weeks after the end of consolidation and for 30 days after the end of treatment
Arm/Group | Gemcitabine | Gemcitabine + Radiation
Serious Adverse Events (participants affected / at risk) | 28/35 | 28/34
Other Adverse Events (participants affected / at risk) | 5/35 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (N=35) | Gemcitabine + Radiation (N=34)
Anemia (Blood and lymphatic system disorders) | 2 | 6
Leukopenia (Investigations) | 5 | 11
Neutrophenia (Investigations) | 14 | 14
Lymphopenia (Investigations) | 0 | 1
Thrombocytopenia (Investigations) | 2 | 7
Transfusion: platelets (Blood and lymphatic system disorders) | 0 | 1
Transfusion:PRBCS (Blood and lymphatic system disorders) | 2 | 6
Cardiac-Ischemia (Cardiac disorders) | 1 | 0
Edema (General disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Thrombosis/Embolism (Vascular disorders) | 1 | 0
Fatigue (General disorders) | 2 | 11
Weight loss (Investigations) | 0 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 6
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 10
Vomiting (Gastrointestinal disorders) | 3 | 9
Diarrhea W/O prior colostomy (Gastrointestinal disorders) | 1 | 2
Melena/GI bleeding (Gastrointestinal disorders) | 0 | 2
Alkaline phosphatase increased (Investigations) | 1 | 2
Bilirubin increased (Metabolism and nutrition disorders) | 1 | 1
Gamma-glutamyl transpeptidase (GGT) increase (Investigations) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3
AST increased (Hepatobiliary disorders) | 1 | 0
ALT increased (Hepatobiliary disorders) | 1 | 1
Infection W/grade 3 or 4 neutropenia (Infections and infestations) | 1 | 1
Infection with unknown ANC (Infections and infestations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Abonominal pain (Gastrointestinal disorders) | 0 | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Plumonary-other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (N=35) | Gemcitabine + Radiation (N=34)
Anemia (Blood and lymphatic system disorders) | 4 | 1
Weight loss (General disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No